CLINICAL TRIAL: NCT03259555
Title: A Multicenter, Randomized, Double-blind Trial of Brexpiprazole Versus Placebo for the Acute Treatment of Manic Episodes, With or Without Mixed Features, Associated With Bipolar I Disorder
Brief Title: A Trial to Assess Brexpiprazole Versus Placebo for the Treatment of Acute Manic Episodes Associated With Bipolar I Disorder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 331-201-00080
Record Dates: First submitted 2017-08-04; First posted 2017-08-23 (Actual); Results first posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Bipolar I Disorder; Manic Episode
Keywords: Brexpiprazole; Bipolar; Manic episode
MeSH Terms: conditions — Mania | interventions — brexpiprazole

STUDY DESIGN:
Intervention Model Description: Participants received a dose of brexpiprazole or placebo for a maximum of 21 days and were evaluated throughout the duration of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Brexpiprazole (Experimental): Participants received a starting dose of 2 milligrams (mg)/day brexpiprazole from Days 1 to 3, followed by titration to 3 mg/day on Day 4. Participants may have been titrated (or re-titrated) to a higher dose of brexpiprazole, up to a maximum of 4 mg/day, based on treatment response and at the investigator's discretion anytime at Day 7 or thereafter. Participants who were unable to tolerate their current dose could have been titrated down to a minimum of 2 mg/day any time after Day 4.
  Interventions: Drug: Brexpiprazole
- Placebo (Placebo Comparator): Matching placebo was administered in the same way as brexpiprazole to maintain the blind.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Brexpiprazole — Brexpiprazole was administered orally with flexible dosing from 2 to 4 mg/day; titrated to a maximum of 4 mg/day for 3 weeks.
  Arms: Brexpiprazole
Drug: Placebo — Administered orally daily for 3 weeks.
  Arms: Placebo

SUMMARY:
To demonstrate the efficacy of brexpiprazole for the acute treatment of manic episodes, with or without mixed features, in participants with a diagnosis of bipolar I disorder.

DETAILED DESCRIPTION:
A multicenter, randomized, double-blind trial of brexpiprazole versus placebo for the acute treatment of manic episodes, with or without mixed features, associated with bipolar I disorder. This study also demonstrated the safety and tolerability of brexpiprazole in the study population of males and females aged 18 to 65 years (inclusive, at time of consent).

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants, ages 18 to 65 years, inclusive, at the time of informed consent.
* Participants willing to discontinue all prohibited medications to meet protocol-required washouts prior to and during the trial period.
* Participants with a Diagnostic & Statistical Manual on Mental Disorders, 5th Edition (DSM-5) diagnosis of bipolar I disorder displaying an acute manic episode with or without mixed features requiring hospitalization. Diagnosis confirmed by the MINI International Neuropsychiatric Interview and a history of at least 1 previous manic episode with or without mixed features with manic symptoms of sufficient severity to require one of the following interventions: hospitalization or treatment with a mood stabilizer, or treatment with an antipsychotic agent. "Require" was defined as an intervention that occurred rather than one that was recommended.
* Young-mania rating scale (YMRS) score of ≥24 at screening and baseline.

Exclusion Criteria:

* Sexually active male or women of childbearing potential who did not agree to practice 2 different methods of birth control or remain abstinent during the trial and for 30 days after the last dose of investigational medicinal product.
* Females who were breastfeeding and/or who had a positive pregnancy test result prior to receiving trial medication.
* Participants considered unresponsive to clozapine or who were only responsive to clozapine.
* Participants with a history of DSM-5 diagnosis other than bipolar I disorder, including schizophrenia, schizoaffective disorder, major depressive disorder, attention-deficit/hyperactivity disorder, delirium, dementia, amnestic, or other cognitive disorders. Also, participants with borderline, paranoid, histrionic, schizotypal, schizoid, or antisocial personality disorder. All other current diagnoses must have been discussed with the medical monitor.
* Participants whose current manic episode had lasted for more than 4 weeks overall, or who had required hospitalization >21 days for the current acute episode at the time of the screening visit, excluding hospitalization for psychosocial reasons.
* Participant with manic symptoms better accounted for by another general medical condition or direct physiological effect of substance (for example, medication).
* Participants who have had electroconvulsive treatment within the past 2 months.
* Participants with a positive drug screen for cocaine or other illicit drugs.
* Abnormal laboratory test results, vital signs or electrocardiogram findings, unless based on investigator's judgment the findings are not medically significant or would not impact the safety of the participant or the interpretation of the trial results.
* Rapid cyclers with more than 6 episodes in the previous year.
* Participants with hypothyroidism or hyperthyroidism (unless condition has been stabilized with medications for at least the past 90 days) or an abnormal result for free thyroxine at screening.
* Participants with uncontrolled hypertension or symptomatic hypotension or orthostatic hypotension.
* Participant with epilepsy or history of seizures.
* Participants who participated in a clinical trial within the last 60 days or who participated in more than 2 clinical trials within the past year.
* Use of psychotropic medications (other than benzodiazepines) within 7 days of the baseline YMRS.
* Participants who currently had clinically significant neurological, hepatic, renal, metabolic, hematological, immunological, cardiovascular, pulmonary, or gastrointestinal disorders.
* Participants who received brexpiprazole in any prior clinical trial or currently taking commercially available brexpiprazole (Rexulti).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2017-09-14 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Leoni, M.D., Study Director — Otsuka Pharmaceutical Development & Commercialization, Inc.
Locations (48):
- United States (29):
  - Woodland International Research Group, Little Rock, Arkansas
  - Woodland Research Northwest, LLC, Rogers, Arkansas
  - ProScience Research Group, Culver City, California
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Behavioral Research Specialists, LLC, Glendale, California
  - Pacific Research Partners, LLC, Oakland, California
  - NRC Research Institute, Orange, California
  - Asclepes Research Centers, Panorama City, California
  - Ci Trials, Riverside, California
  - Sharp Vista Hospital, San Diego, California
  - Galiz Research, Hialeah, Florida
  - Advanced Research Institute of Miami, Homestead, Florida
  - Florida Behavioral Medicine, Largo, Florida
  - Optimus U Corporation, Miami, Florida
  - Behavioral Clinical Research, Inc., North Miami, Florida
  - Segal Trials, North Miami, Florida
  - Radiant Research Inc., Atlanta, Georgia
  - Alexian Brothers Center for Psychiatric Research, Hoffman Estates, Illinois
  - CBH Health, Gaithersburg, Maryland
  - Advanced Clinical Research Center, LLC, St Louis, Missouri
  - Richard H Weisler, MD, PA, and Associates, Raleigh, North Carolina
  - SP Research PLLC, Oklahoma City, Oklahoma
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - Carolina Clinical Trials, Inc., Charleston, South Carolina
  - University of Texas at Austin, Austin, Texas
  - Community Clinical Research, Inc., Austin, Texas
  - Pillar Clinical Research, LLC, Garland, Texas
  - Pillar Clinical Research, LLC, Richardson, Texas
  - Mid Columbia Research, Richland, Washington
- Bulgaria (9):
  - Mental Health Center Prof. Dr. Ivan Temkov - Burgas EOOD, Burgas
  - State Psychiatry Hospital - Kardzhali, Kardzhali
  - State Psychiatry Hospital Sv. Ivan Rilski, Novi Iskar
  - University Multiprofile Hospital for Active Treatment Sveti Georgi EAD, Plovdiv
  - Mental Health Center - Ruse EOOD, Rousse
  - University Multiprofile Hospital for Active Treatment Alexandrovska EAD, Sofia
  - Multiprofile Hospital for Active Treatment - Targovishte AD, Targovishte
  - Mental Health Center - Veliko Tarnovo EOOD, Veliko Tarnovo
  - Mental Health Center - Vratsa EOOD, Vratsa
- Poland (4):
  - Samodzielny Publiczny Psychiatryczny Zaklad Opieki Zdrowotnej im. Dr. Stanislawa Deresza w Choroszczy, Choroszcz
  - Uniwersyteckie Centrum Kliniczne w Gdansku Klinika Psychiatrii Doroslych, Gdansk
  - NZOZ Centrum Medyczne HCP Sp. z o. o., Poznan
  - NZOZ Prywatna Klinika Psychiatryczna Inventiva, Tuszyn
- Serbia (6):
  - Clinic for Psychiatric Disorders Dr Laza Lazarevic, Belgrade
  - Clinical Center of Serbia, Belgrade
  - Clinical Hospital Center Dr Dragisa Misovic-Dedinje, Belgrade
  - Special Hospital for Psychiatric Diseases Kovin, Kovin
  - Clinical Center Kragujevac, Kragujevac
  - Clinical Center of Vojvodina, Novi Sad

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The trial population consisted of adult participants (18 to 65 years) diagnosed with bipolar I disorder displaying an acute manic episode with or without mixed features requiring hospitalization.
Groups:
- Brexpiprazole: Brexpiprazole was administered orally with flexible dosing from 2 to 4 milligrams (mg)/day; titrated to a maximum of 4 mg/day.
- Placebo: Matching placebo was administered orally in the same way as brexpiprazole to maintain the blind.
Period: Overall Study
Arm/Group | Brexpiprazole | Placebo
Started | 158 | 164
Received At Least 1 Dose of Study Drug (Randomized participants who received at least 1 dose of study drug were analyzed for safety.) | 158 | 163
Completed | 124 | 134
Not Completed | 34 | 30
Not completed — Adverse Event | 6 | 4
Not completed — Lack of Efficacy | 6 | 4
Not completed — Lost to Follow-up | 0 | 2
Not completed — Non-Compliance With Study Drug | 1 | 0
Not completed — Progressive Disease | 0 | 2
Not completed — Withdrawal by Subject | 19 | 16
Not completed — Physician Decision | 1 | 2
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline population consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Brexpiprazole | Placebo | Total
Number analyzed (Participants) | 158 | 164 | 322
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.4 (11.7) | 44.5 (11.2) | 44.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 83 | 163
  Male | 78 | 81 | 159
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 16 | 22 | 38
  Not Hispanic or Latino | 141 | 141 | 282
  Unknown | 0 | 1 | 1
  Ethnicity - Other | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 95 | 113 | 208
  Black or African American | 54 | 51 | 105
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Race - Other | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline In Young-Mania Rating Scale (YMRS) Score At Week 3
Description: The YMRS was utilized to assess a participant's level of manic symptoms. It consists of 11 items: 1) elevated mood, 2) increased motor activity-energy, 3) sexual interest, 4) sleep, 5) irritability, 6) speech (rate and amount), 7) language-thought disorder, 8) content, 9) disruptive-aggressive behavior, 10) appearance, and 11) insight. Seven items are rated on a 0- to 4-scale, while four items (Items 5, 6, 8, and 9) are rated on a 0- to 8-scale with 0, 2, 4, 6, and 8 being the possible scores (twice the weight of the other items). For all items, 0 is the "best" rating and the highest score (4 or 8) is the 'worst' rating. The YMRS total score is the sum of ratings for all 11 items; therefore, possible total scores range from 0 to 60, with higher scores signifying more severe manic symptoms. Comparison between treatment groups was carried out using mixed-effect model repeated measure (MMRM).
Time Frame: Baseline, Week 3
Population: Full Analysis Set: all participants who received at least 1 dose of study drug and had a baseline value and at least 1 valid post-randomization efficacy evaluation for YMRS Total Score in the double-blind treatment phase at the specified timepoint.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 124 | 134
units on a scale | -10.6 (0.72) | -10.8 (0.70)
Statistical Analysis 1: Comparison: Brexpiprazole vs Placebo; Test type: Superiority; p = 0.8797, Mixed-effect Model Repeated Measure; An "unstructured" covariance was used; Treatment difference = 0.14, 95% CI 2-sided [-1.74 to 2.03] — Comparison between treatment groups was carried out using MMRM, with study center, treatment group, visit, and treatment group-by-visit interaction as factor and baseline-by-visit interaction as a covariate. An "unstructured" covariance was used

2. Secondary Outcome: Change From Baseline In Clinical Global Impression-Bipolar (CGI-BP) Severity Score In Mania At Week 3
Description: The CGI-BP scale refers to the global impression of the participant with respect to bipolar disorder. The scale rates the participant's severity of illness (CGI-BP severity of illness: mania, depression, and overall bipolar illness) based on a 7-point scale: 1 = normal, not at all ill, 2 = minimally ill, 3 = mildly ill, 4 = moderately ill, 5 = markedly ill, 6 = severely ill, 7 = very severely ill.
Time Frame: Baseline, Week 3
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Brexpiprazole | Placebo
Number analyzed (Participants) | 124 | 134
units on a scale | -1.12 (1.06) | -1.21 (1.13)

ADVERSE EVENTS:
Time Frame: From Day 1 (after dosing) through 6 weeks (3 weeks treatment, 3 weeks safety follow-up).
Arm/Group | Brexpiprazole | Placebo
All-Cause Mortality (participants affected / at risk) | 0/158 | 0/163
Serious Adverse Events (participants affected / at risk) | 4/158 | 1/163
Other Adverse Events (participants affected / at risk) | 20/158 | 24/163
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brexpiprazole (N=158) | Placebo (N=163)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Varicella (Infections and infestations) | 1 (1) | 0 (0)
Akathisia (Nervous system disorders) | 1 (1) | 0 (0)
Dystonia (Nervous system disorders) | 1 (1) | 0 (0)
Mania (Psychiatric disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Brexpiprazole (N=158) | Placebo (N=163)
Akathisia (Nervous system disorders) | 8 (8) | 2 (2)
Headache (Nervous system disorders) | 6 (8) | 11 (11)
Constipation (Gastrointestinal disorders) | 2 (2) | 6 (6)
Nausea (Gastrointestinal disorders) | 4 (4) | 5 (6)
Agitation (Psychiatric disorders) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right to review results publications prior to public release and can delay such publications for a period greater than 60 days but no more than 120 days from the date that the publication is submitted to the Sponsor for review. Sponsor can require changes to the publication to protect Sponsor's intellectual property rights and/or confidential information and reserves the right to limit publication timing and scope of data published based on the number of study locations.

DOCUMENTS (2):
  • Study Protocol (2017-12-21): https://cdn.clinicaltrials.gov/large-docs/55/NCT03259555/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-11): https://cdn.clinicaltrials.gov/large-docs/55/NCT03259555/SAP_001.pdf